Official Title: Adapting an Advocacy Services Intervention for Latinx Families of Transitionaged Youth With Autism Spectrum Disorder

NCT Number: NCT06207149

Document Date: 8/25/23 (date of most recent approval by the human subjects protection review board)

Statistical Analysis Plan: First, we will determine whether there are any missing data and impute as needed following Harrell's guidelines (2000). Then, we will determine whether there are demographic differences between the intervention and control groups; we will control for relevant differences, as needed. For the first research question, we will conduct a MANOVA to discern differences in the post scores on knowledge of adult disability services, advocacy skills and comfort, individual advocacy activities, and the Family Empowerment Scale. For the second research question, we will conduct a repeated measures ANOVA by condition. The dependent variables will be the number of services received and unmet service needs.